CLINICAL TRIAL: NCT06772324
Title: An Exploratory Clinical Study of a Low-dose Buprenorphine Patch for the Treatment of Autism Spectrum Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Collaborators: Ping An-Shionogi Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Qingjiu Cao, Chief Physician, Professor, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PKUH6PSCN001
Record Dates: First submitted 2024-12-27; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder
Keywords: low-dose Buprenorphine patch; autism spectrum disorders; Buprenorphine
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: This was a randomized, three-arm, parallel, double-masked study in male/female subjects with ASD with a treatment duration of 56 days. No crossing will be implemented.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization and Masking will be performed via a non-blinded data management team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Very-low dose group (Experimental): Dosing will begin on Day 1, and the buprenorphine transdermal patch will be changed every 7 days, i.e., Day 8, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50, and Day 57. Of these, Day 15, Day 22, Day 36, Day 43, and Day 50 will require subjects and their guardians to self-replace the patch at home. Day 1, Day 8, Day 29, and Day 57 will receive medication in the hospital.
  Day1 0 mg patch; all subjects receiving their medication in-hospital after completing all tests assessed at baseline; Day8, Day29 one-ninth of a 5mg patch and replaced with a 0mg patch before returning home from the test; all subjects will receive medication upon arrival at the hospital before completing relevant assessment tests; Day57 one-ninth of a 5-mg patch; all subjects will receive medication upon arrival at the hospital before completing relevant assessment tests and will be allowed to go home only after removing the used buprenorphine transdermal patch at the end of the assessment;
  Interventions: Drug: NORSPAN Buprenorphine Transdermal Patchs for Very-low dose group
- Lower dose group (Experimental): Dosing will begin on Day 1, and the buprenorphine transdermal patch will be changed every 7 days, i.e., Day 8, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50, and Day 57. Of these, Day 15, Day 22, Day 36, Day 43, and Day 50 will require subjects and their guardians to self-replace the patch at home. Day 1, 8, 29, and 57 will receive medication in the hospital.
  Day1 one-ninth of a 5 mg patch; all subjects receiving their medication in-hospital after completing all tests assessed at baseline; Day8, Day29 one-ninth of a 5mg patch and replaced with one-ninth of a new 5mg patch before returning home from the test; all subjects will receive medication upon arrival at the hospital before completing relevant assessment tests; Day57 one-ninth of a 5-mg patch; all subjects will receive medication upon arrival at the hospital before completing relevant assessment tests and will be allowed to go home only after removing the used buprenorphine transdermal patch at the end of the assessment;
  Interventions: Drug: NORSPAN Buprenorphine Transdermal Patchs for Lower dose group
- Higher dose group (Experimental): Dosing will begin on Day 1, and the buprenorphine transdermal patch will be changed every 7 days, i.e., Day 8, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50, and Day 57. Of these, Day 15, Day 22, Day 36, Day 43, and Day 50 will require subjects and their guardians to self-replace the patch at home. Day 1, 8, 29, and 57 will receive medication in the hospital.
  Day1 one-third of a 5 mg patch; all subjects receiving their medication in-hospital after completing all tests assessed at baseline; Day8, Day29 one-third of a 5mg patch wil be replaced with one-third of a new 5mg patch before returning home from the test; all subjects will receive medication upon arrival at the hospital before completing relevant assessment tests; Day57 one-third of a 5-mg patch; all subjects will receive medication upon arrival at the hospital before completing relevant assessment tests and will be allowed to go home only after removing the used buprenorphine transdermal patch at the end of the assessment;
  Interventions: Drug: NORSPAN Buprenorphine Transdermal Patchs for higher dose group

INTERVENTIONS:
Drug: NORSPAN Buprenorphine Transdermal Patchs for Very-low dose group — Very-low dose group will receive medication on arrival before completing the relevant assessment tests; the very-low dose group will be administered 1/9 of a 5mg buprenorphine transdermal patch and replaced with a 0mg patch before returning home from the examination.
  Arms: Very-low dose group
Drug: NORSPAN Buprenorphine Transdermal Patchs for Lower dose group — The lower dose group will be administered 1/9 of a 5mg buprenorphine transdermal patch.
  Arms: Lower dose group
Drug: NORSPAN Buprenorphine Transdermal Patchs for higher dose group — The higher dose group will be administered 1/3 of a 5mg buprenorphine transdermal patch.
  Arms: Higher dose group

SUMMARY:
This study evaluates the safety and efficacy of low-dose buprenorphine in patients with ASD by using standard ASD symptom assessment methods (e.g., SRS-2 and ABC) as well as AI-assisted analyses utilizing exploratory gaze patterns in conjunction with fMRI and electroencephalogram measurements to assess changes in brain functional status.

DETAILED DESCRIPTION:
The study aims to assess the safety and efficacy of buprenorphine in patients with autism spectrum disorders (ASD) in very low, lower, and higher dose groups and to explore the sensitivity and specificity of ophthalmoscopy for evaluating the efficacy of ASD treatment. Combined neuroimaging techniques to examine the effects of buprenorphine on neurologic function in ASD.

In this study, changes in functional brain status will be assessed by using standard ASD symptom assessment methods (e.g., SRS and ABC) as well as algorithms utilizing AI's exploratory gaze patterns in conjunction with functional magnetic resonance and electroencephalography imaging to evaluate changes in the functional brain state of the very low-dose group (5 mg 1/9 at follow-up only), the lower-dose group (5 mg 1/9/week) and the higher-dose group (5 mg 1/3/week) buprenorphine safety and efficacy in patients with ASD. This study will validate the results of previous studies based on humans and rodents and is expected to develop an effective drug for treating the core symptoms of ASD with significant social and economic benefits.

This is a randomized, three-arm, double-blind study in male/female subjects with ASD with a treatment duration of 56 days. Items to be evaluated include efficacy on ASD symptoms, safety, Day57's buprenorphine drug concentration in plasma, and changes in oculomotor, functional magnetic resonance, and electroencephalographic data before and after treatment. The effective dose is estimated based on the results of preclinical studies of buprenorphine in ASD model mice, using a dose of one-third or one-ninth of the available 5-mg buprenorphine transdermal patch.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male/female;
* Age:6-18 years at the time of randomization;
* Clinical diagnosis in accordance with the DSM-5 diagnosis of ASD;
* Diagnosis of ASD using the K-SADS-PL-C DSM-5 and CARS;
* A severity score of ≥ 4 on the CGI scale;
* Subjects must be able to participate and deemed suitable for participation in the study, at the investigator's discretion, and be able to follow the study evaluation schedule;
* The parent or guardian agrees to accompany the subject to all clinical visits and to provide information about the subject's behavior and symptoms, and must agree to supervise the subject's compliance with protocol-specified procedures and the use of study drug doses;
* The parent or guardian is willing and able to give written informed consent in accordance with local requirements. When the subject is capable of making the decision to consent to participation in the study, the subject is likewise willing and able to provide written informed consent in accordance with local requirements.

Exclusion Criteria:

1. Neurologic/Psychiatric Disorders

   * Concurrent comorbidity with any other mental disorder (other than ADHD) as diagnosed by the K-SADS-PL-C DSM-5;
   * Neurologic disorders or prior head trauma resulting in coma;
   * Unstable or uncontrollable clinically significant psychiatric and/or neurological disorders that may interfere with safety or efficacy outcome;
   * Unstable or uncontrolled irritability in the judgment of the investigator;
   * Any suicide attempts in the opinion of the investigator at the time of screening that he/she is at risk for suicidal behavior or in his/her medical history;
   * A history of seizures within the past 6 months;
   * A history of alcohol or other substance abuse/dependence.
2. Cardiovascular Disease

   * Current cardiovascular disease not effectively controlled in the opinion of the investigator;
   * Clinically significant abnormalities (e.g., twice consecutive measurements) as confirmed by ECG at screening, including, but not limited to: QTc: ≥450 milliseconds, absence of predominant sinus rhythm, and second or third degree a-v block.
3. Diseases of other organ systems

   * Accompanying other diseases or conditions (pulmonary, gastrointestinal, hepatic, renal, metabolic, immune system, or obesity) that may interfere or whose treatment may interfere with the conduct of the study; or where, in the opinion of the Investigator, discontinuation of the Prohibited Substance may pose an unacceptable risk to the subject.
   * Evidence of gastrointestinal bleeding, e.g., active gastric ulcer;
   * History of coagulopathy, bleeding disorders or blood disorders;
4. Other exclusion criteria

   * Marked respiratory depression;
   * Acute or severe bronchial asthma;
   * Known or suspected paralytic bowel obstruction;
   * Allergic to buprenorphine;
   * Participation in a drug study within 30 days prior to randomization or within 5 times the half-life of the molecule to be studied, whichever is longer; or drug study; or participation in a study testing a medical device within 30 days prior to randomization, or the device is still in action. active;
   * History of blood loss greater than 250 mL within 3 months prior to screening;
   * Medications permitted since 4 weeks prior to screening that have NOT been clearified and stable, and medications permitted for the treatment of epilepsy since 3 months prior to screening that have NOT been clearified and stable.
   * Usage of a prohibited medication within 2 weeks prior to the screening visit (and ensuring at least 4 weeks of washout time prior to the baseline assessment) or usage of a prohibited medication within 5 times of half-life prior to the randomization (whichever is longer).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness Scale (SRS) | screening period, Day 1, Day 29, Day 57.
  It is a screening tool for the diagnosis and assessment of autism in children aged 4-18 years that recognizes the presence of ASD-related social impairments and quantifies their severity. It identifies ASD-related social impairments and quantifies their severity. The scale consists of 65 questions categorized as Social Self-Consciousness, Social Cognition, Social Communication, and Social Self-Expression. The scale consists of 65 questions divided into five dimensions: social awareness, social cognition, social communication, social motivation, and autistic behavior.
  There are a total of 65 questions, with a minimum score of 1 and a maximum score of 4 for each question, with a total score range of 65-260.
  The higher the score, the more significant the condition.
Autism Behavior Checklist （ABC） | Day 1, Day 29, Day 57.
  It is a behavioral assessment tool for children with autism and is primarily used to assess the outcome of patients with mental retardation and autism. The scale consists of 58 items divided into 5 factors: emotional lability/self-injurious aggression (15 items), social withdrawal/stagnation (16 items), stereotypic behavior (7 items), hyperactivity (16 items), and inappropriate speech (4 items).
  There are a total of 58 questions, each with a minimum score of 0 and a maximum score of 3, with a total score range of 0-174. The higher the score, the more significant the condition.

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | screening period, Day 1, Day 29, Day 57.
  It is an overall rating scale that is applicable to any psychiatric treatment and research subject.
  The comprehensive score is based on the two dimensions of efficacy and adverse reactions. The most effective and least adverse reaction score is 1 point, while the least effective and most adverse reaction score is 16 points. The score range is 1-16.
Treatment Emergent Symptom Scale (TESS) | Day8, Day 29, Day 57.
  It is a medication safety evaluation tool used by psychiatrists to assess side effects in patients taking psychotropic medications.
  There are a total of 29 questions, each with three dimensions: severity, relationship with medication, and treatment. The score range for severity is 0-4, with higher scores indicating greater severity. The score range for the relationship with drugs is 0-4, and the higher the score, the greater the relationship with drugs. The processing range is 0-6, and the higher the score, the greater the degree of processing.
Patient Global Impression (PGI) | Day 1, Day 29, Day 57.
  There are two questions in total, namely severity and overall evaluation of efficacy. The score range for severity is 0-4, with higher scores indicating greater severity. The score range for the overall efficacy evaluation is 0-7, with higher scores indicating greater deterioration of the condition.
Eye Tracking Test | screening period, Day 1, Day8, Day 29, Day 57.
  Subjects will be seated in front of a monitor equipped with eye-tracking equipment. The equipment will be adjusted according to the subject's actual condition before the formal start. After commissioning, a 1-2 minute video will be played and eye movement data will be collected during the video.
  The eye movement data will be analyzed by quantifying the ratio of the length of time the patient looks at the face of the person appearing in the video to the length of time he/she looks at the geometric figure, the length of time he/she looks at the eye region of the person, and so on.
functional magnetic resonance imaging (fMRI) | screening period, Day 57.
  Includes resting-state fMRI data, DTI data, and ASL data, collected during the screening period and at visit 5, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Sixth Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided